CLINICAL TRIAL: NCT06720350
Title: Efficacy of Romosozumab and Denosumab Combined Treatment in Postmenopausal Osteoporosis Patients with Multiple Fragility Fractures
Acronym: MORD
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: MAROP.ROM.DEN
Record Dates: First submitted 2024-12-03; First posted 2024-12-06 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Osteoporosis in Post-menopausal Women
Keywords: Osteoporosis; Combination Therapy; Romosozumab; Denosumab
MeSH Terms: conditions — Osteoporosis | interventions — romosozumab; Denosumab

STUDY DESIGN:
Intervention Model Description: Each of treatment options will randomized in patients with postmenopausal women.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Romosozumab and denosumab combination (Experimental): Romosozumab 210 mg subcutaneously per month combined with denosumab 60mg subcutaneously per 6 months
  Interventions: Drug: Romosozumab and Denosumab Combination Therapy
- Romosozumab (Active Comparator): Romosozumab 210 mg subcutaneously per month
  Interventions: Drug: Romosozumab Prefilled Syringe [Evenity]
- Denosumab (Active Comparator): denosumab 60mg subcutaneously per 6 months
  Interventions: Drug: Denosumab (Prolia)

INTERVENTIONS:
Drug: Romosozumab and Denosumab Combination Therapy — Romosozumab 210mg per month and denosumab 60mg per 6 months will be applied
  Arms: Romosozumab and denosumab combination
Drug: Romosozumab Prefilled Syringe [Evenity] — Romosozumab 210mg subcutaneously per month
  Arms: Romosozumab
Drug: Denosumab (Prolia) — Denosumab 60 mg subcutaneously per 6 months
  Arms: Denosumab

SUMMARY:
The aim of this clinical trial is to investigate the effectiveness of romosozumab started without stopping denosumab in patients diagnosed with postmenopausal osteoporosis with a very high risk of fragility fractures and who is under at least 2 years of denosumab treatment. The main questions aimed to answer are:

* Does it effective to prevent fractures add Romosozumab to ongoing denosumab treatment?
* If it is appropiate to quit denosumab for starting 1 year romosozumab treatment?
* If there is complications in denosumab and romosozumab combination treatment?

Researchers will compare the Romosozumab 210mg subcutaneous(sc) monthly plus denosumab 60mg per 6 months sc treatment to prooceeding denosumab treatment and romosozumab 210mg monthly treatment in patient whom denosumab cessaced.

Participians are postmenopousal women with osteoporosis and they are under at least 2 years of treatment with denosumab and they will:

* Add 210 mg monthly romosozumab sc injection or switch to 210 mg monthly romosozumab sc injection or proceed 60mg per 6 months denosumab sc injection
* Visit the clinic at least once every 3 months and first month of new treatment regimen, blood tests per 3 months and Bone mineral density examination per 6 months
* Keep a diary of their symptoms

DETAILED DESCRIPTION:
Osteoporosis, whether accompanied by low bone resorption, microarchitectural deterioration, and fragility, leads to poor bone strength and increased risk of fracture. Decreased bone strength can also be due to external factors including bone formation and resorption (turnover), bone geometry (bone size and shape), and bone mineral density (BMD), including microarchitecture. Osteoporotic fractures lead to a significant decrease in quality of life with increased morbidity, mortality, and disability. More than 50 percent of postmenopausal white women will have an osteoporotic fracture, and only 33 percent of older women with a hip fracture are able to live independently.

The World Health Organization (WHO) has defined diagnostic thresholds for low bone density and osteoporosis based on measurements of bone density versus the young adult reference (T score). Postmenopausal women with osteoporosis have decreased bone loss and/or experienced associated bone loss.

Romosozumab is a drug used to treat osteoporosis. Romosozumab is an FDA-cleared humanized monoclonal antibody sclerostin inhibitor used to treat postmenopausal osteoporosis at high risk of fracture, including patients with a history of osteoporotic fractures, those who have failed or are tolerant to other available osteoporosis therapies, and those who have failed or are tolerant to other available osteoporosis therapies. It increases bone formation and impairs bone resorption.

For most postmenopausal women with osteoporosis, oral bisphosphonates are preferred as initial therapy because of their efficacy, affordability, and availability of long-term safety data. Treatment selection should be based on efficacy, safety, cost, freedom, and the individual's fracture risk.

In a 2019 meta-analysis of 107 studies evaluating pharmacological treatments in postmenopausal women with osteoporosis, alendronate, zoledronic acid, risdronate, denosumab, romosozumab, and estrogen with progestin were found to reduce the risk of hip fractures. Alendronate, zoledronic acid, rosedronate, ibandronate, denosumab, abaloparatide, teriparatide, parathyroid hormone (1.84), romosozumab, raloxifene, bazedoxifene, lasofoxifene, estrogen with progestin, tibolone, and calcitonin were found to reduce the risk of vertebral fractures. Anabolic agents (teriparatide, abaloparatide, romosozumab) and denosumab were found to have the highest relative efficacy, but few studies compared the drugs in terms of fracture prevention.

Current evidence suggests that Romosozumab therapy is a good option for osteoporosis in postmenopausal women with a history of multiple fractures and BMD measurements below L1-L4 or Femoral Neck T-scores below -3.5. The anabolic agent romosozumab uniquely stimulates bone formation and inhibits bone resorption. In postmenopausal women at very high risk of fracture, literature data suggests that anabolic therapies prevent fractures to a greater extent compared with oral bisphosphonates. Romosozumab induces a greater BMD response than abaloparatide or teriparatide, but clinical experience is limited and long-term side effects are uncertain.

In Lancet's systematic review of osteoporosis treatment, it was recommended that long-term follow-up, fracture outcome studies be conducted to evaluate the effectiveness of combined treatments in patients with high fracture risk.

Combination therapies refer to the sequential or simultaneous administration of two drugs. In the previous ARCH study, a better treatment response was seen in the group given 70mg/week alendronate after 12 months of 210mg/month romosozumab treatment compared to the group given 70mg/week alendronate alone. In the FRAME study, new fractures were significantly less in the group given 12 months of 60mg/6month denosumab after 12 months of 210mg/month romosozumab treatment compared to the group given 12 months of 60mg/6month denosumab after 12 months of placebo. These two studies were phase 3 studies that demonstrated the efficacy of sequential therapies and romosozumab in the treatment of osteoporosis.

In the DATA-Switch study published in Lancet in 2015, which evaluated the combination and sequential treatments of teriparatide and denosumab, 3 groups were formed with a total of 48 months of sequential 24-month treatments, and these groups were given Denosumab after Teriparatide; Teriparatide after Denosumab and Denosumab after the combination of these two drugs. The results of the study showed that teriparatide after denosumab did not prevent sufficient fracture risk and did not provide sufficient improvement in BMD measurements, in line with the literature. In addition, the use of denosumab was found to be more appropriate both after combined treatment and after teriparatide alone. The best BMD improvement was determined in the group that received denosumab after combined treatment.

In a study conducted by McClung et al., the study included patients who were in the placebo group in the first 24 months of the Romosozumab Phase 2 study (NCT00896532) and were randomized to placebo or denosumab for the next 12 months. In this phase 2 study, 210 mg/month romosozumab was finally administered to all study arms. The study results showed that romosozumab at least maintains BMD improvement after denosumab, while it is more effective in naïve patients. The STRUCTURE phase 2 extension study also showed that romosozumab provided minimal BMD improvement in the patient group who received a second course of 12-month romosozumab treatment after denosumab. In this context, it is possible to say that romosozumab is more effective in naive patients, but this situation brings to mind the problem that like the use of teriparatide alone after denosumab is not appropriate the use of romosozumab after denosumab may decrease its effectiveness, and may not be appropriate in terms of effectiveness and cost, even if it does not worsen the disease. IIn a case written by Kashii et al. in 2020, the patient who applied after missing his follow-up for 3 months had 9 months since his last denosumab dose at the time of application. Although there was no new fracture development, the patient was switched to romosozumab treatment because sufficient BMD improvement could not be detected with denosumab. The patient, who did not have back pain complaints at the time of the transition and in the 1st month, had back pain complaints at the 3rd month follow-up, but no fracture was detected in the direct radiography performed on the patient and MRI could not be performed due to the patient's claustrophobia. In the direct radiography taken in the 4th month of romosozumab, a total of 5 new fractures at the thoracic and lumbar levels were detected. Although romosozumab treatment was completed in the 6th month of this case, sufficient improvement was not detected in BMD measurements. In a case written by Krikelis et al., denosumab was stopped and romosozumab was started in a patient who developed 1 vertebral fracture under denosumab. 5 new thoracic and lumbar vertebral fractures were detected in the 6th month of romosozumab treatment. This situation was attributed to the withdrawal effect of denosumab, and romosozumab was discontinued and denosumab was started again. After 1 month, the patient's back pain regressed. At this point, due to insufficient literature, they considered adding denosumab again while continuing romosozumab, but they could not do it. Two published cases in this treatment regimen and literature data on the use of teriparatide after denosumab show us that the effect of adding romosozumab should be investigated while continuing denosumab treatment, especially in patients with a high risk of rebound-related vertebral fractures, when anabolic agent treatment is planned.

In a study conducted by Adami et al., which is the only example in the literature on combined treatment with Romosozumab and Denosumab, romosozumab was started in drug-naive patients in the first of the 3 study arms, romosozumab was added to the group that had been using denosumab for over 2 years in the second group, and denosumab treatment was continued alone in the last group. After 6 months of follow-up, romosozumab administered to naive patients was found to be superior to other treatments in reducing the risk of hip fractures, while similar results were found with combined treatment in reducing the risk of lumbar fractures. IIn the group where denosumab was continued alone, the reduction in fracture risk was found to be significantly less than in the other groups. This study did not include information on side effects and complications.

It is obvious that there is a lack of information in the literature on the treatment arrangement without stopping denosumab in patients diagnosed with postmenopausal osteoporosis with a very high risk of fragility fractures, when it is planned to switch to romosozumab after denosumab. At this point, a study should be planned on this subject. The aim of our study is to investigate the effectiveness of romosozumab, which is started without stopping denosumab, and therefore the effectiveness of romosozumab-denosumab combined treatment in patients with postmenopausal osteoporosis diagnosed with a very high risk of fragility fractures and receiving denosumab treatment.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal Women
* Patients with Osteoporosis
* Patients aged between 55 and 85 years old

Exclusion Criteria:

* Patient with history of Serebrovascular diseases
* Patient with history of Miyocardial Infarction
* Patients who have calcium metabiolism disturbances
* Patients with chronic kidney diseases
* Patient with history of allergic reactions to denosumab or romosozumab

Ages: 55 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Postmenopausal women aged 55-85 years old
Enrollment: 60 (Estimated)
Dates: Start 2025-01-15 (Estimated); Primary Completion 2026-10-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
New Fracture | 1 year and 9 months
  If the patient exposed new fracture along treatment period
Bone Mineral Density | 1 year
  Bone mineral density before treatment regimen and after treatment done

SECONDARY OUTCOMES:
New fracture at long term follow up | 5 years
  If the patient exposed new fracture along long term follow up (Phase 2 of this study) period
Beta Crosslaps | 6 months interval
  Beta Crosslaps value througout treatment regimen per 6 months interval

CONTACTS AND LOCATIONS:
Overall Officials: Canan Sanal, Associate Profesor, Study Director — Marmara University Medical School
Locations (1):
- Marmara University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Adami G, Pedrollo E, Rossini M, Fassio A, Braga V, Pasetto E, Pollastri F, Benini C, Viapiana O, Gatti D. Romosozumab added to ongoing denosumab in postmenopausal osteoporosis, a prospective observational study. JBMR Plus. 2024 Feb 7;8(4):ziae016. doi: 10.1093/jbmrpl/ziae016. eCollection 2024 Apr. PMID 38544922
- [Background] Krikelis M, Gazi S, Trovas G, Makris K, Chronopoulos E, Tournis S. Progression of multiple vertebral fractures after denosumab discontinuation under treatment with romosozumab. A case-report. Joint Bone Spine. 2024 Sep;91(5):105754. doi: 10.1016/j.jbspin.2024.105754. Epub 2024 Jun 26. PMID 38942353
- [Background] Kashii M, Ebina K, Kitaguchi K, Yoshikawa H. Romosozumab was not effective in preventing multiple spontaneous clinical vertebral fractures after denosumab discontinuation: A case report. Bone Rep. 2020 Jun 5;13:100288. doi: 10.1016/j.bonr.2020.100288. eCollection 2020 Dec. PMID 32548215
- [Background] Langdahl BL, Libanati C, Crittenden DB, Bolognese MA, Brown JP, Daizadeh NS, Dokoupilova E, Engelke K, Finkelstein JS, Genant HK, Goemaere S, Hyldstrup L, Jodar-Gimeno E, Keaveny TM, Kendler D, Lakatos P, Maddox J, Malouf J, Massari FE, Molina JF, Ulla MR, Grauer A. Romosozumab (sclerostin monoclonal antibody) versus teriparatide in postmenopausal women with osteoporosis transitioning from oral bisphosphonate therapy: a randomised, open-label, phase 3 trial. Lancet. 2017 Sep 30;390(10102):1585-1594. doi: 10.1016/S0140-6736(17)31613-6. Epub 2017 Jul 26. PMID 28755782
- [Background] McClung MR, Bolognese MA, Brown JP, Reginster JY, Langdahl BL, Shi Y, Timoshanko J, Libanati C, Chines A, Oates MK. Skeletal responses to romosozumab after 12 months of denosumab. JBMR Plus. 2021 Jun 3;5(7):e10512. doi: 10.1002/jbm4.10512. eCollection 2021 Jul. PMID 34258507
- [Background] Leder BZ, Tsai JN, Uihlein AV, Wallace PM, Lee H, Neer RM, Burnett-Bowie SA. Denosumab and teriparatide transitions in postmenopausal osteoporosis (the DATA-Switch study): extension of a randomised controlled trial. Lancet. 2015 Sep 19;386(9999):1147-55. doi: 10.1016/S0140-6736(15)61120-5. Epub 2015 Jul 2. PMID 26144908
- [Background] Brown JP, Engelke K, Keaveny TM, Chines A, Chapurlat R, Foldes AJ, Nogues X, Civitelli R, De Villiers T, Massari F, Zerbini CAF, Wang Z, Oates MK, Recknor C, Libanati C. Romosozumab improves lumbar spine bone mass and bone strength parameters relative to alendronate in postmenopausal women: results from the Active-Controlled Fracture Study in Postmenopausal Women With Osteoporosis at High Risk (ARCH) trial. J Bone Miner Res. 2021 Nov;36(11):2139-2152. doi: 10.1002/jbmr.4409. Epub 2021 Aug 10. PMID 34190361
- [Background] Reid IR, Billington EO. Drug therapy for osteoporosis in older adults. Lancet. 2022 Mar 12;399(10329):1080-1092. doi: 10.1016/S0140-6736(21)02646-5. PMID 35279261
- [Background] Shoback D, Rosen CJ, Black DM, Cheung AM, Murad MH, Eastell R. Pharmacological Management of Osteoporosis in Postmenopausal Women: An Endocrine Society Guideline Update. J Clin Endocrinol Metab. 2020 Mar 1;105(3):dgaa048. doi: 10.1210/clinem/dgaa048. PMID 32068863
- [Background] Saag KG, Petersen J, Brandi ML, Karaplis AC, Lorentzon M, Thomas T, Maddox J, Fan M, Meisner PD, Grauer A. Romosozumab or Alendronate for Fracture Prevention in Women with Osteoporosis. N Engl J Med. 2017 Oct 12;377(15):1417-1427. doi: 10.1056/NEJMoa1708322. Epub 2017 Sep 11. PMID 28892457
- [Background] Kendler DL, Marin F, Zerbini CAF, Russo LA, Greenspan SL, Zikan V, Bagur A, Malouf-Sierra J, Lakatos P, Fahrleitner-Pammer A, Lespessailles E, Minisola S, Body JJ, Geusens P, Moricke R, Lopez-Romero P. Effects of teriparatide and risedronate on new fractures in post-menopausal women with severe osteoporosis (VERO): a multicentre, double-blind, double-dummy, randomised controlled trial. Lancet. 2018 Jan 20;391(10117):230-240. doi: 10.1016/S0140-6736(17)32137-2. Epub 2017 Nov 9. PMID 29129436
- [Background] Barrionuevo P, Kapoor E, Asi N, Alahdab F, Mohammed K, Benkhadra K, Almasri J, Farah W, Sarigianni M, Muthusamy K, Al Nofal A, Haydour Q, Wang Z, Murad MH. Efficacy of Pharmacological Therapies for the Prevention of Fractures in Postmenopausal Women: A Network Meta-Analysis. J Clin Endocrinol Metab. 2019 May 1;104(5):1623-1630. doi: 10.1210/jc.2019-00192. PMID 30907957
- [Background] Ayers C, Kansagara D, Lazur B, Fu R, Kwon A, Harrod C. Effectiveness and Safety of Treatments to Prevent Fractures in People With Low Bone Mass or Primary Osteoporosis: A Living Systematic Review and Network Meta-analysis for the American College of Physicians. Ann Intern Med. 2023 Feb;176(2):182-195. doi: 10.7326/M22-0684. Epub 2023 Jan 3. PMID 36592455
- [Background] Viswanathan M, Reddy S, Berkman N, Cullen K, Middleton JC, Nicholson WK, Kahwati LC. Screening to Prevent Osteoporotic Fractures: Updated Evidence Report and Systematic Review for the US Preventive Services Task Force. JAMA. 2018 Jun 26;319(24):2532-2551. doi: 10.1001/jama.2018.6537. PMID 29946734
- [Background] Eastell R, Rosen CJ, Black DM, Cheung AM, Murad MH, Shoback D. Pharmacological Management of Osteoporosis in Postmenopausal Women: An Endocrine Society* Clinical Practice Guideline. J Clin Endocrinol Metab. 2019 May 1;104(5):1595-1622. doi: 10.1210/jc.2019-00221. PMID 30907953
- [Background] Porter JL, Varacallo MA. Osteoporosis(Archived). 2023 Aug 4. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK441901/ PMID 28722930
- [Background] Singh S, Dutta S, Khasbage S, Kumar T, Sachin J, Sharma J, Varthya SB. A systematic review and meta-analysis of efficacy and safety of Romosozumab in postmenopausal osteoporosis. Osteoporos Int. 2022 Jan;33(1):1-12. doi: 10.1007/s00198-021-06095-y. Epub 2021 Aug 25. PMID 34432115
- [Background] Cosman F, Crittenden DB, Adachi JD, Binkley N, Czerwinski E, Ferrari S, Hofbauer LC, Lau E, Lewiecki EM, Miyauchi A, Zerbini CA, Milmont CE, Chen L, Maddox J, Meisner PD, Libanati C, Grauer A. Romosozumab Treatment in Postmenopausal Women with Osteoporosis. N Engl J Med. 2016 Oct 20;375(16):1532-1543. doi: 10.1056/NEJMoa1607948. Epub 2016 Sep 18. PMID 27641143